CLINICAL TRIAL: NCT00263861
Title: Impact of Treatment With Taxane or Platinum-Containing Regimens on Peripheral Nerve Functioning in Older Cancer Patients With Diabetes: An Exploratory Study
Brief Title: Nerve Function in Older Diabetic Patients Who Are Undergoing Chemotherapy for Metastatic Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Constance Visovsky, PhD, RN, ACNP, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CWRU6Z03; P30CA043703 (NIH); CASE-CWRU-6Z03 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: management of therapy complications — Patients undergo an interview and clinical evaluation to measure demographic data, cutaneous sensation, gait and balance, vibration, lower extremity muscle strength, orthostatic blood pressure, and glycemic control.

SUMMARY:
RATIONALE: Learning about the side effects of chemotherapy may help plan treatment and may help patients live more comfortably.

PURPOSE: This clinical trial is studying nerve function in older diabetic patients who are undergoing chemotherapy for metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine changes in peripheral nerve function in older patients with diabetes and metastatic solid tumors treated with taxane or platinum-containing chemotherapy regimens.
* Determine the extent to which age, pre-existing diabetes mellitus, and level of glycemic control predict a differential pattern in outcome beyond the effect of the drugs in patients treated with these regimens.
* Develop a clinical assessment that would predict whether or not patients with diabetes mellitus are more or less susceptible to the neurotoxic effects of chemotherapy.

OUTLINE: This is a longitudinal study.

Patients undergo an interview and clinical evaluation to measure demographic data, cutaneous sensation, gait and balance, vibration, lower extremity muscle strength, orthostatic blood pressure, and glycemic control. Patients are evaluated at baseline, every 3 weeks during chemotherapy for up to 4 treatments, and at 2 months after completion of treatment.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor

  * Metastatic disease (stage IV)
* Planning neoadjuvant or adjuvant treatment of locoregional definitive or systemic therapy comprising ≥ 1 of the following:

  * Taxane (paclitaxel or docetaxel)
  * Platinum (cisplatin, carboplatin, or oxaliplatin)
* Diagnosis of type I or II diabetes mellitus

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other disease that reduces peripheral nerve function (e.g., HIV/AIDS, uremia, spinal injuries, alcoholism, or CNS problems)

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy
* No prior or concurrent neurotoxic drugs (i.e., vincristine)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cutaneous sensation as measured by Semmes-Weinstein monofilaments | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment
Gait and balance as measured by Tinetti Performance Oriented Assessment of Gait and Balance Instrument | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment
Vibration as measured by tuning fork | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment
Lower extremity muscle strength as measured by Dynamometer | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment
Blood pressure changes | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment
Glycemic control as measured by Glycosylated Hemoglobin Assay | baseline, every 3 weeks for 4 courses, and then 2 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Constance Visovsky, PhD, RN, ACNP, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States